CLINICAL TRIAL: NCT02244411
Title: Exercise and QUality Diet After Leukemia: The EQUAL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Johns Hopkins University (Other); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-164
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Adult Survivors of Childhood Leukemia
Keywords: EQUAL; Exercise; Diet; Physical activity; 14-164
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires; Weights and Measures; Waist Circumference; Blood Pressure

ARMS (2):
- Intervention group (Experimental): Participants will be assigned an individual diet & physical activity counselor through Healthways at Hopkins. This counselor will stay with the participant for the 24 months. The primary communication with the counselor will be via website & email. Participants will be encouraged to consume a low-calorie, low-salt diet with 7-12 daily servings of fruits, vegetables & low-fat dairy products. Calorie goals are based upon weight at study entry & whether or not the weight loss goal has been met. Participants will gradually build to ≥ 180 minutes of moderate to vigorous physical activity per week, using the activity of their own choosing & gradually adding bouts of ≥ 10 minutes in length. Monitoring & Counselor Contacts: the first 3 months, the participants are encouraged to log into the web hub on a daily basis to record weight, food intake, & physical activity. Participants who decline or drop out of the intervention program will remain on-study doing home visits & questionnaires.
  Interventions: Behavioral: individual diet & physical activity counselor and website through Healthways at Hopkins; Behavioral: questionnaires; Other: fasting blood draw, measurement of height, weight and waist circumference, and blood pressure
- control group (Active Comparator): Participants will receive general information brochures on healthy living and weight loss but will not have access to the Healthways at Hopkins website or counselors.
  Interventions: Behavioral: self directed weight loss; Behavioral: questionnaires; Other: fasting blood draw, measurement of height, weight and waist circumference, and blood pressure

INTERVENTIONS:
Behavioral: individual diet & physical activity counselor and website through Healthways at Hopkins — Phone and web-based weight loss intervention (via Healthways at Hopkins counselor and website) focused on increasing physical activity and adhering to a healthy diet. Participants will log diet, physical activity, and weight in web-hub. Counselors will have access to this information to direct participants to goals and achievements.
  Arms: Intervention group
Behavioral: self directed weight loss — Participants will be given information and links to CDC and American Cancer Society recommendations for healthy eating and physical activity.
  Arms: control group
Behavioral: questionnaires — Participants will complete behavioral questionnaires as well as diet and physical activity assessments through CCSS-based study website as baseline, 12 and 24 months.
Other: fasting blood draw, measurement of height, weight and waist circumference, and blood pressure — During three time periods, at baseline and at 12 and 24 months.

SUMMARY:
The EQUAL study has been designed for adult survivors of childhood acute lymphoblastic leukemia (ALL) who are overweight or obese. The purpose of this study is to see if diet and exercise can help people lose weight and improve other health problems. This two year study will compare two methods of informing participants about ways to lose weight.

ELIGIBILITY:
Inclusion Criteria:

Eligibility will be confirmed via the CCSS-based medical record and by a series of questions on the EQUAL website, prior to consent.

* Participation in the CCSS cohort
* Diagnosed with acute lymphoblastic leukemia < 18 years of age
* Cancer free at time of study enrollment
* Current age ≥ 18 years
* A body mass index (BMI) ≥ 25 kg/m2 (overweight or obese), as determined by self-reported height and weight on the most recent CCSS questionnaire
* Internet access and a personal email account
* Able to read and comprehend informed consent

Exclusion Criteria:

* Prior history of congestive heart failure, coronary artery disease, myocardial infarction, stroke, or unstable angina;
* Medical condition for which weight loss might be contraindicated or which would cause weight loss, such as pregnancy, anorexia or bulimia;
* Use of prescription weight loss medication within the previous 6 months
* History of total body irradiation (TBI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Weight loss | 24 months
  Weight loss will be evaluated in an intent-to-treat analysis with a linear mixed effects model with robust standard errors and an unstructured covariance matrix(50) using weight measured at each time points (0, 12 months and 24 months after randomization) as the outcome modeled as a function of time, randomization arm, a history of CRT, gender, age, and race together with interaction terms between time and randomization arm.

CONTACTS AND LOCATIONS:
Overall Officials: Chaya Moskowitz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/